CLINICAL TRIAL: NCT01877252
Title: National Registry Investigating the Effectiveness of Different First-line Treatment Strategies in Patients With Critical Limb Ischemia
Brief Title: Registry of First-line Treatments in Patients With Critical Limb Ischemia
Acronym: CRITISCH
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Collaborators: Deutsches Institut für Gefäßmedizinische Gesundheitsforschung gGmbH (DIGG) (Unknown); Deutsche Gesellschaft für Gefäßchirurgie und Gefäßmedizin (Unknown)
Responsible Party: Principal Investigator, Dr. Theodosios Bisdas, Dr. med., St. Franziskus Hospital
Other Study IDs: CRITISCH132105
Record Dates: First submitted 2013-05-20; First posted 2013-06-13 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Critical Limb Ischemia
Keywords: critical limb ischemia; endovascular treatment; open surgical repair; diabetic foot
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetic Foot | interventions — Polytetrafluoroethylene; Polyethylene Terephthalates; Angioplasty, Balloon; Stents; Drug-Eluting Stents; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Endovascular treatment: Angioplasty +/- stent
  Interventions: Procedure: Endovascular revascularization
- Open treatment: Bypass (vein or prosthetic)
  Interventions: Procedure: Surgical revascularization
- Patchplasty/Hybrid treatment: Femoral artery patchplasty +/- profundoplasty +/- endovascular treatment
  Interventions: Procedure: Surgical revascularization; Procedure: Endovascular revascularization
- Conservative treatment: no vascular intervention
  Interventions: Other: No vascular intervention

INTERVENTIONS:
Procedure: Surgical revascularization
  Other Names: Vein; PTFE; Dacron; Femoral artery patchplasty; Profunda patchplasty
  Groups: Open treatment; Patchplasty/Hybrid treatment
Procedure: Endovascular revascularization
  Other Names: Balloon angioplasty; Stent; Drug-eluting balloon; Drug-eluting stent; Lysis
  Groups: Endovascular treatment; Patchplasty/Hybrid treatment
Other: No vascular intervention
  Other Names: Major amputation; Minor amputation; Sympatholysis; Conservative treatment
  Groups: Conservative treatment

SUMMARY:
The principal research question is which treatment modality between open surgical, endovascular and conservative therapy is the most effective in terms of limb salvage, survival and reinterventions in patients with critical limb ischemia

DETAILED DESCRIPTION:
The target population consists of patients suffering from critical limb ischemia (CLI) lasting more than 2 weeks. CLI is defined as rest pain or tissue loss (Fontaine stages III-IV or Rutherford classes 4 to 6) and/or ankle-brachial index < 0.40. Patient with acute limb-threatening ischemia, bone fractures in the relevant areas, nonatherosclerotic disease (e.g. arteriitis) and documented hypercoagulable diseases will be excluded from this study. There will be no experimental or control groups. The comparison groups will be:

Group 1: Best endovascular treatment (angioplasty +/- stent) Group 2: Best surgical treatment [bypass (vein or prosthetic)] Group 3: Femoral artery patchplasty +/- profundoplasty (+/- endovascular treatment) Group 4: Best conservative treatment

The proposed sample size amounts to 1200 patients.

To be assessed for eligibility (n=1200) To be allocated to trial (n=1000) To be analysed (n=900)

In CRITISCH registry, randomization or blinding is not feasible, because optimized standard care will be performed as established at each participating centre (best medical treatment). Data storage, validation, monitoring, update, backup and analysis will be performed centrally following established procedures. Web-based software will be used to develop a data model representing the data structure. The data validation will include standard data validation techniques such as the manual review of selected variables and the routine check of missing and outlying data points. Regional staff will be instructed and supervised by study nurse, who will perform the study monitoring. Assessment of relevant prognostic factors during the statistical analysis will prevent biased results due to the non-randomized design and the potential structural inequality.

ELIGIBILITY:
Inclusion Criteria:

* Rest pain or tissue loss (Fontaine stages III-IV or Rutherford classes 4 to 6) and/or ankle-brachial index < 0.40

Exclusion Criteria:

* Acute limb-threatening ischemia
* Bone fractures in the relevant areas
* Non-atherosclerotic disease (e.g. arteriitis)
* Documented hypercoagulable diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of patients suffering from critical limb ischemia lasting more than 2 weeks
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Amputation-free survival | at 2 years
  Above-ankle amputation of the index limb or death (any cause), whichever occurred first

SECONDARY OUTCOMES:
Perioperative death | 30 days
Major adverse limb event (MALE) | at 1 year, at 2 years
  above ankle amputation of the index limb or major intervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis)
Major adverse cardiovascular event (MACCE) | at 30 days, at 1 year, at 2 years
  myocardial infarction, stroke or death (any cause)
Sustained clinical improvement | at 1 year, at 2 years
  upward shift on the Rutherford or Fontaine classification to a level of intermittent claudication in amputation-free surviving patients without the need for repeated target lesion revascularization (TLR) (primary improvement) or after repeated TLR (secondary improvement)
Hemodynamic failure | at 30 days, at 1 year, at 2 years
  first occurrence of any of the following events in a time-to-event fashion: (a) major amputation (transtibial or above) and/or (b) reintervention to maintain vascular patency in the index limb and/or (c) failure to increase ankle-brachial-index (ABI) by at least 0.15 postprocedure] and/or (d) decrease in ABI by 0.15

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Surgery, St. Franziskus Hospital, Münster, Germany

REFERENCES:
- [Background] Setacci C, de Donato G, Teraa M, Moll FL, Ricco JB, Becker F, Robert-Ebadi H, Cao P, Eckstein HH, De Rango P, Diehm N, Schmidli J, Dick F, Davies AH, Lepantalo M, Apelqvist J. Chapter IV: Treatment of critical limb ischaemia. Eur J Vasc Endovasc Surg. 2011 Dec;42 Suppl 2:S43-59. doi: 10.1016/S1078-5884(11)60014-2. PMID 22172473
- [Background] Becker F, Robert-Ebadi H, Ricco JB, Setacci C, Cao P, de Donato G, Eckstein HH, De Rango P, Diehm N, Schmidli J, Teraa M, Moll FL, Dick F, Davies AH, Lepantalo M, Apelqvist J. Chapter I: Definitions, epidemiology, clinical presentation and prognosis. Eur J Vasc Endovasc Surg. 2011 Dec;42 Suppl 2:S4-12. doi: 10.1016/S1078-5884(11)60009-9. PMID 22172472
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Bradbury AW, Adam DJ, Bell J, Forbes JF, Fowkes FG, Gillespie I, Ruckley CV, Raab GM; BASIL trial Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: An intention-to-treat analysis of amputation-free and overall survival in patients randomized to a bypass surgery-first or a balloon angioplasty-first revascularization strategy. J Vasc Surg. 2010 May;51(5 Suppl):5S-17S. doi: 10.1016/j.jvs.2010.01.073. PMID 20435258
- [Background] Conte MS, Geraghty PJ, Bradbury AW, Hevelone ND, Lipsitz SR, Moneta GL, Nehler MR, Powell RJ, Sidawy AN. Suggested objective performance goals and clinical trial design for evaluating catheter-based treatment of critical limb ischemia. J Vasc Surg. 2009 Dec;50(6):1462-73.e1-3. doi: 10.1016/j.jvs.2009.09.044. Epub 2009 Nov 7. PMID 19897335
- [Derived] Stavroulakis K, Borowski M, Torsello G, Bisdas T; CRITISCH Collaborators. One-Year Results of First-Line Treatment Strategies in Patients With Critical Limb Ischemia (CRITISCH Registry). J Endovasc Ther. 2018 Jun;25(3):320-329. doi: 10.1177/1526602818771383. Epub 2018 Apr 26. PMID 29968501
- [Derived] Meyer A, Fiessler C, Stavroulakis K, Torsello G, Bisdas T, Lang W; CRITISCH collaborators. Outcomes of dialysis patients with critical limb ischemia after revascularization compared with patients with normal renal function. J Vasc Surg. 2018 Sep;68(3):822-829.e1. doi: 10.1016/j.jvs.2017.12.048. Epub 2018 Mar 26. PMID 29598891
- [Derived] Stavroulakis K, Borowski M, Torsello G, Bisdas T; CRITISCH collaborators. Association between statin therapy and amputation-free survival in patients with critical limb ischemia in the CRITISCH registry. J Vasc Surg. 2017 Nov;66(5):1534-1542. doi: 10.1016/j.jvs.2017.05.115. Epub 2017 Aug 12. PMID 28807382
- [Derived] Uhl C, Steinbauer M, Torsello G, Bisdas T; The CRITISCH collaborators. Outcomes After Endovascular Revascularization in Octogenarians and Non-Octogenarians With Critical Limb Ischemia. J Endovasc Ther. 2017 Aug 1;24(4):471-477. doi: 10.1177/1526602817711424. Epub 2017 Jun 5. PMID 28578624
- [Derived] Bisdas T, Borowski M, Stavroulakis K, Torsello G; CRITISCH Collaborators. Endovascular Therapy Versus Bypass Surgery as First-Line Treatment Strategies for Critical Limb Ischemia: Results of the Interim Analysis of the CRITISCH Registry. JACC Cardiovasc Interv. 2016 Dec 26;9(24):2557-2565. doi: 10.1016/j.jcin.2016.09.039. PMID 28007205
- [Derived] Meyer A, Lang W, Borowski M, Torsello G, Bisdas T; CRITISCH collaborators. In-hospital outcomes in patients with critical limb ischemia and end-stage renal disease after revascularization. J Vasc Surg. 2016 Apr;63(4):966-73. doi: 10.1016/j.jvs.2015.10.009. Epub 2016 Feb 1. PMID 26843355
- [Derived] Bisdas T, Borowski M, Torsello G; First-Line Treatments in Patients With Critical Limb Ischemia (CRITISCH) Collaborators. Current practice of first-line treatment strategies in patients with critical limb ischemia. J Vasc Surg. 2015 Oct;62(4):965-973.e3. doi: 10.1016/j.jvs.2015.04.441. Epub 2015 Jul 14. PMID 26187290
- See also: German Society for Vascular Surgery and Medicine — http://www.gefaesschirurgie.de